CLINICAL TRIAL: NCT04305132
Title: Can Electroconvulsive Therapy Alter Retinal Nerve Fiber Layer Thickness of Patients With Depression
Brief Title: Effect of Electroconvulsive Therapy on Retinal Nerve Fiber Layer Thickness in Depression
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Mehmet Diyaddin Güleken (Other)
Responsible Party: Sponsor-Investigator, Mehmet Diyaddin Güleken, MDGuleken, Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital
Organization: Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital (Other)
Other Study IDs: MDGuleken
Record Dates: First submitted 2020-03-09; First posted 2020-03-12 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Depression
Keywords: depression; electroconvulsive therapy; retinal nerve fiber layer; optical coherence tomography
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- Depression: Subjects with depression treated with electroconvulsive therapy
  Interventions: Device: Electroconvulsive therapy
- Healthy: Healthy subjects

INTERVENTIONS:
Device: Electroconvulsive therapy — Thymatron System IV electroconvulsive therapy device
  Groups: Depression

SUMMARY:
The aim of this study is to investigate the changes in the retinal nerve fiber layer thickness of the patients with depression who received electroconvulsive therapy by means of optical coherence tomography.

DETAILED DESCRIPTION:
Major depression (MD) is a mood disorder that is common in the society, has negative effects on emotion, thought and behavior, and leads to significant impairments in functionality. Electroconvulsive therapy (ECT) is a highly effective and reliable biological treatment method used in psychiatric diseases for a long time. The most common use in psychiatry is depression. Studies have shown that ECT causes a broadly distributed increase in brain gray matter volume (especially the temporal lobe) in MD patients. Optical coherence tomography (OCT) is a non-invasive medical imaging method that displays biological tissue layers by taking high resolution tomographic sections. Alterations in the thickness of the retinal nerve fiber layer (RNFL), which is a layer of the ganglion cell complex in the retina of the eye and consists of ganglion cell axons, occur due to axonal damage in the retinal nerve tissue. Since RNFL is in a similar form with the brain gray matter tissue, recently, neurological and psychiatric studies have been conducted to provide data regarding the neurodegeneration occurring in the brain tissue. In the study, it is aimed to assess the possible cortical volume changes of patients by measuring changes in the retinal layers due to ECT in patients with depression. In other words, considering that ECT causes an increase in brain volume, it is to observe whether this increase is reflected in the retinal nerve fiber layer thickness.

ELIGIBILITY:
Inclusion Criteria:

* Subject diagnosed as unipolar depression
* Subject with depression to be treated with electroconvulsive therapy
* Subject with depression having a Standardized Mini Mental Test score of >23

Exclusion Criteria:

* Any comorbid psychiatric condition (including alcohol / substance use)
* Having any major neurological (i.e.: cerebrovascular disease, multiple sclerosis, etc.) disease
* Having any major medical (i.e.: diabetes mellitus, myocardial infarction, etc.) disease
* History of or having any ocular trauma, disease or surgery, any retinal disease, refraction defect
* To be treated with electroconvulsive therapy in the last 6 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will include 25 volunteered inpatient or outpatient subjects with depression diagnosed with Structured Clinical Interview for DSM 5 Clinical Version (SCID 5/CV) who are followed-up at the Sağlık Bilimleri Üniversitesi Gazi Yaşargil Training and Research Hospital and 25 healthy volunteers matched with these patients in terms of age and gender. In order to measure the severity of the disease, subjects with depression will be administered Hamilton Depression Rating Scale (HAM-D), Young Mania Rating Scale (YMRS) and Clinical Global Impression Scale (CGI) before ECT, after the first ECT session and after the last ECT last session. The Symptom Check List-90-Revised (SCL-90-R) will be administered to healthy volunteers after enrollment.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Changes of retinal nerve fiber layer thickness | About 4 weeks
  Changes of retinal nerve fiber layer thickness of subjects with depression before and after electroconvulsive therapy

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet D Güleken, MD, Study Director — Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital
Locations (1):
- Sağlık Bilimleri Üniversitesi Gazi Yaşargil Tranining and Research Hospital, Diyarbakır, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available with six months of study completion.
Access Criteria: Data access requests will be reviewed by an independent reviewer. Requestors will be required to sign a Data Access Agreement.

REFERENCES:
- [Background] Gazdag G, Ungvari GS. Electroconvulsive therapy: 80 years old and still going strong. World J Psychiatry. 2019 Jan 4;9(1):1-6. doi: 10.5498/wjp.v9.i1.1. eCollection 2019 Jan 4. PMID 30631748
- [Background] Ousdal OT, Argyelan M, Narr KL, Abbott C, Wade B, Vandenbulcke M, Urretavizcaya M, Tendolkar I, Takamiya A, Stek ML, Soriano-Mas C, Redlich R, Paulson OB, Oudega ML, Opel N, Nordanskog P, Kishimoto T, Kampe R, Jorgensen A, Hanson LG, Hamilton JP, Espinoza R, Emsell L, van Eijndhoven P, Dols A, Dannlowski U, Cardoner N, Bouckaert F, Anand A, Bartsch H, Kessler U, Oedegaard KJ, Dale AM, Oltedal L; GEMRIC. Brain Changes Induced by Electroconvulsive Therapy Are Broadly Distributed. Biol Psychiatry. 2020 Mar 1;87(5):451-461. doi: 10.1016/j.biopsych.2019.07.010. Epub 2019 Jul 25. PMID 31561859
- [Background] Pan J, Zhou Y, Xiang Y, Yu J. Retinal nerve fiber layer thickness changes in Schizophrenia: A meta-analysis of case-control studies. Psychiatry Res. 2018 Dec;270:786-791. doi: 10.1016/j.psychres.2018.10.075. Epub 2018 Oct 30. PMID 30551326
- [Background] Mutlu U, Colijn JM, Ikram MA, Bonnemaijer PWM, Licher S, Wolters FJ, Tiemeier H, Koudstaal PJ, Klaver CCW, Ikram MK. Association of Retinal Neurodegeneration on Optical Coherence Tomography With Dementia: A Population-Based Study. JAMA Neurol. 2018 Oct 1;75(10):1256-1263. doi: 10.1001/jamaneurol.2018.1563. PMID 29946702